CLINICAL TRIAL: NCT04548375
Title: Multicenter Outcome Registry of AnaLgesic Effect of SCS(MORALES) Registry Protocol
Status: Recruiting | Type: Observational
Sponsor: Cardio Surgical Partners (Network)
Responsible Party: Sponsor
Other Study IDs: PainReg
Record Dates: First submitted 2020-08-26; First posted 2020-09-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: SCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SCS — Conventional SCS implants approved through all payors(government and private) for FDA approved indications

SUMMARY:
The objective is to provide information to help the physician community decide the most effective type of device/therapy that would work for their patients, based off of the etiology of pain, the location of the pain for sustained pain relief.

DETAILED DESCRIPTION:
This registry will enroll patients that qualify for an SCS implant, for approved pain areas, as defined by medicare guidelines, and follow these patients for up to 12 months for denovo implants. For patients who have lost their pain relief over time, with a prior implanted device, this registry will follow a change out to another vendor/therapy, and follow those patients for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* FDA approved indications for SCS implants, for commercial and government(medicare, medi-cal etc) approved payors

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All SCS implants
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain relief | 12 months
  Percent of patient who show a change in Pain Scale (PIPS) >50% at the end of follow up period of 12 months

OTHER OUTCOMES:
Sustained change of pain over the follow up period | 12 months
  Sustained Percentage change in Pain Scale (PIPS)>50% for the 12 month follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Summit Surgery Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No